CLINICAL TRIAL: NCT06516068
Title: A Multicenter, Randomized, Open-label Phase II Clinical Study on the Efficacy and Safety of HRS-1893 in Obstructive Hypertrophic Cardiomyopathy Subjects.
Brief Title: A Trial of HRS-1893 in Patients With Obstructive Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1893-201
Record Dates: First submitted 2024-06-28; First posted 2024-07-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1893 (Experimental)
  Interventions: Drug: HRS-1893

INTERVENTIONS:
Drug: HRS-1893 — HRS-1893

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HRS-1893 for obstructive hypertrophic cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old, gender unlimited;
2. The diagnosis was obstructive hypertrophic cardiomyopathy.
3. Echocardiographic laboratory tests showed LVEF≥60%;
4. No previous left ventricular systolic dysfunction at any time (LVEF < 45%);
5. Understand the study procedure and sign the informed consent in person, willing to strictly follow the clinical study protocol to complete the study.

Exclusion Criteria:

1. Known or suspected invasive, genetic or storage diseases (e.g. Noonan syndrome, Fabre's disease, amyloidosis) that cause cardiac hypertrophy (similar to oHCM);
2. Previous left ventricular systolic dysfunction at any time in the clinical course (LVEF < 45%);
3. Previous history of aortic stenosis or subaortic fixed stenosis;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-11 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The subjects' left ventricular outflow tract pressure gradient (Valsalva LVOT-G) was assessed for changes from the baseline after performing the Valsalva maneuver | After 12 weeks of HRS-1893 treatment

SECONDARY OUTCOMES:
Change in peak oxygen uptake (pVO2) and carbon dioxide ventilation equivalent (VE/VCO2) | Baseline to Week 12
Change in LVEF | Baseline to Week 12
Change in LVOT-VTI | Baseline to Week 12
Change in LV-FS | Baseline to Week 12
Change in LV-GLS | Baseline to Week 12
Change in Rest LVOT-G | Baseline to Week 12
Change in Valsalva LVOT-G | Baseline to Week 12
Change in cardiac troponin | Baseline to Week 12
Change in NT-proBNP | Baseline to Week 12
Change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) | Baseline to Week 12
Proportion of participants with ≥ 1 class improvement in NYHA Functional Class | Baseline to Week 12
Incidence and severity of any adverse events (AESI, SAE, TRAE, TEAE) | Through study completion, an average of 68 weeks
plasma concentration of HRS-1893 | Through study completion, an average of 68 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences (CAMS), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided